CLINICAL TRIAL: NCT03124446
Title: Mindfulness-Based College: Stage 1 Randomized Controlled Trial for Emerging Adult Well-Being
Brief Title: Mindfulness-Based College: Stage 1
Acronym: MB-College
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1608001570
Record Dates: First submitted 2017-04-14; First posted 2017-04-21 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Diet Habit; Physical Activity; Sleep; Loneliness; Emotional Regulation; Alcohol Consumption, Youth; Stress, Psychological
Keywords: mindfulness, meditation, emerging adults, young adults, undergraduate students, stress, health
MeSH Terms: conditions — Feeding Behavior; Motor Activity; Emotional Regulation; Underage Drinking; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Overall, a superiority randomized controlled trial with parallel groups will be performed with 30 participants per arm. Participants will be randomly assigned to MB-College or enhanced usual care control.
Masking Description: Data analysts will be blinded to treatment allocation and randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based College (Experimental): MB-College is an 8-week, 9-session curriculum providing systematic and intensive training in mindfulness meditation practices, applied to health behaviors relevant to college students. The curriculum is based on the manualized and standardized Mindfulness-Based Stress Reduction. The course builds a foundation of mindfulness self-regulation skills, including attention control, self-awareness and emotion regulation. It then directs those skills towards participants' relationships with health-related factors particularly salient in college undergraduates, including physical activity, diet, alcohol consumption, sleep, stress, social relationships, cognitive performance, and emotion regulation. Health behavior goal setting, and support for behavior change are integrated in the curriculum.
  Interventions: Behavioral: Mindfulness-Based College
- Enhanced Usual Care Control (Active Comparator): Participants in the enhanced usual care control group were spoken with by trained study staff, and as part of the enhanced usual care, were offered a referral to the study's psychiatrist and University counseling resources, if anxiety, depression, or suicidal ideation levels at baseline or follow-up reached clinical levels on the Beck Anxiety Inventory or the Revised Centers for Epidemiologic Studies Depression (CESD-R) scale. Participants in the control group were eligible to take the MB-College program during the following university term.
  Interventions: Behavioral: Enhanced Usual Care Control

INTERVENTIONS:
Behavioral: Mindfulness-Based College — MB-College is an 8-week, 9-session curriculum providing systematic and intensive training in mindfulness meditation practices, applied to health behaviors relevant to college students. The curriculum is based on the manualized and standardized Mindfulness-Based Stress Reduction. The course builds a foundation of mindfulness self-regulation skills, including attention control, self-awareness and emotion regulation. It then directs those skills towards participants' relationships with health-related factors particularly salient in college undergraduates, including physical activity, diet, alcohol consumption, sleep, stress, social relationships, cognitive performance, and emotion regulation. Health behavior goal setting, and support for behavior change are integrated in the curriculum.
  Arms: Mindfulness-Based College
Behavioral: Enhanced Usual Care Control — Participants in the enhanced usual care control group were spoken with by trained study staff, and as part of the enhanced usual care, were offered a referral to the study's psychiatrist and University counseling resources, if anxiety, depression, or suicidal ideation levels at baseline or follow-up reached clinical levels on the Beck Anxiety Inventory or the Revised Centers for Epidemiologic Studies Depression (CESD-R) scale. Participants in the control group were eligible to take the MB-College program during the following university term.
  Arms: Enhanced Usual Care Control

SUMMARY:
Mindfulness interventions are increasingly offered to undergraduate students at universities world-wide, however the evidence base is very limited. The objective is to evaluate effects of a customized mindfulness intervention (called Mindfulness-Based College) on undergraduate student health. A superiority randomized controlled trial with parallel groups will be performed with 30 participants in each arm. Participants will be randomly assigned to Mindfulness-Based College or health education waitlist control. Investigators will be blinded to treatment allocation. Participants will be assessed at baseline, 10 weeks, and six months. The primary outcome is a college health summary score, including seven evidence-based determinants of health particularly relevant to college student well-being: body mass index, physical activity, diet, alcohol consumption, sleep quantity, perceived stress, and loneliness. Primary intention-to-treat analyses will evaluate whether MB-College vs. control is associated with the summary score, utilizing generalized linear models. Secondary analyses will evaluate which, if any, of the seven determinants of health are driving associations.

DETAILED DESCRIPTION:
1. Background and Rationale

   Mindfulness interventions in school- and work-place settings are expanding exponentially, often with a limited evidence base. Increasingly, mindfulness interventions are customized to specific populations and health outcomes to increase intervention efficacy and efficiency. Emerging adulthood and the college undergraduate experience is a sensitive life course period, with strong peer effects, diminished parental influence, and compelling opportunities for exploring health behaviors having sustained effects, including social relationships, sleep patterns, alcohol and substance use, dietary patterns, and physical or sedentary activities.6 Few mindfulness interventions focus specifically on this population, but preliminary results are promising. Specifically, a randomized controlled trial (RCT) evaluating effects of the low time-burden Koru mindfulness intervention showed significant improvements in perceived stress, sleep, mindfulness and self-compassion immediately following the 4-week intervention, vs. waitlist control. An intensive mindfulness intervention RCT, customized to enhance physical activity, nutrition, sleep, mindfulness, compassion, relationships and well-being, demonstrated significant improvements in physical health, working memory, standardized test performance, mood, self-esteem, self-efficacy mindfulness and life satisfaction vs. control, at 6 weeks follow-up.8 We developed the moderate intensity Mindfulness-Based College (MB-College) intervention, which in a pre/post pilot study showed significant improvements in emotion regulation, diastolic blood pressure, stress, mindfulness and cognitive performance at 8 weeks follow-up (Table 1). Overall, early studies suggest potential benefit for college student health, however these studies require replication, longer term follow-up, and rigorous study designs.
2. Objective

   The primary objective is to perform an RCT to evaluate effects of MB-College vs. health education waitlist control, on a college undergraduate student health summary score at 6 months follow-up.
3. Methods

Overall, a superiority randomized controlled trial with parallel groups will be performed with 40 participants per arm. Participants will be randomly assigned to MB-College or health education waitlist control. Investigators will be blinded to treatment allocation, including staff performing assessments, randomization, and data analyses. Participants will be assessed at baseline, 10 weeks, and 6 months follow-up. Standard CONSORT guidelines will be followed, including trial registration at ClinicalTrials.gov.

The study population inclusion criteria are 18-28 years of age, current undergraduate student at any university, and English communication. Exclusion criteria follow standard recommendations, specifically current regular meditation practice, substance abuse, suicidal ideation, or history of bipolar or psychotic disorders or self-injurious behaviors.

Participants will be recruited using print medium (e.g. recruitment cards and posters distributed throughout campuses), distributing advertisement graphics via social media, and advertisement emails sent to student listservs.

The intervention is MB-College, which is an 8-week, 9-session curriculum providing systematic and intensive training in mindfulness meditation practices, applied to health behaviors relevant to college students. The curriculum (available upon request) is based on the manualized and standardized Mindfulness-Based Stress Reduction (MBSR) developed at the University of Massachusetts Medical School. The course builds a foundation of mindfulness self-regulation skills, including attention control, self-awareness and emotion regulation. It then directs those skills towards participants' relationships with health-related factors particularly salient in college undergraduates, including physical activity, diet, alcohol consumption, sleep, stress, social relationships, cognitive performance, and emotion regulation. Health behavior goal setting, and support for behavior change are integrated in the curriculum.

The control condition is a health education wait list control, which participants will be offered a 30 minute, one-on-one meeting with the MB-College instructor. There, participants will learn about the MB-College curriculum, and have opportunities to share their relationship with common determinants of undergraduate student health and performance, described above. Together, the student and instructor will explore ways the course may assist in shifting these parts of their lives, as they see best. A deliberate relationship will be formed with the instructor.

The primary outcome is a college health summary score, assessed using the following seven evidence-based determinants of health particularly relevant to college student well-being: body mass index (height and weight, directly assessed using standard epidemiologic methods); physical activity (MET minutes and step counts per week, using validated actigraphy and IPAQ - International Physical Activity Questionnaire); diet (mean daily fruit and vegetable consumption, utilizing validated Willet food frequency questionnaire); alcohol consumption (mean drinks per day, via standard questions from Behavioral Risk Factor Surveillance Survey); sleep quantity (mean sleep hours per night, using Pittsburgh Sleep Quality Index); perceived stress (validated Perceived Stress Scale score); and loneliness (validated R-UCLA [University of California Los Angeles] Loneliness Scale score). Specifically, analyses will assess changes in mean Z-scores of college health summary score, using a single mean health summary score across the seven aforementioned college health domains. Secondary analyses will evaluate which of the seven domains are most driving associations. Further primary analyses will determine if participant-identified health domains to focus on showed improvements in MB-College vs. control, utilizing the z-score approach described above, but restricting only to health domains identified by participants as having high readiness to change.

Secondary outcomes, utilizing the National Institutes of Health (NIH) Science of Behavior Change Framework and NIH Stage Model for Intervention Development, include measures of self-regulation hypothesized to be proximal targets to the mindfulness intervention such as self-awareness (e.g. via validated Multidimensional Assessment of Interoceptive Awareness) and attention control (e.g. via validated Sustained Attention to Response Task and Mindful Attention Awareness Scale). Potential effect modifiers assessed include age, race, ethnicity, and socioeconomic status, as well as adverse childhood experiences utilizing the Adverse Childhood Experiences Questionnaire.

All in-person assessments will take place at the Brown School of Public Health by trained research staff experienced in assessing all aforementioned measures. For the estimated timeline, please see Figure 1.

Stratified randomization will be used for intervention allocation, performed using Research Randomizer (www.randomizer.org). Variables used to create strata include gender and race/ethnicity. Blinded, simple random sampling will occur within each strata.

The analytic approach will evaluate whether MB-College vs. control is associated with college health summary score, described above. Analyses will incorporate generalized linear models (GLM) with properly chosen link functions, performed using generalized estimating equations (GEE) with robust standard error estimators. Following "intention-to-treat" principles, analyses will be conducted on all participants, regardless of intervention completion.

Focus groups of participants will take place following MB-College, facilitated by Prof. Abigail Harrison, who is an experienced focus group moderator and researcher. The goal is to customize MB-College to the unique needs of this population. NVivo software (QSR International, Burlington, MA) will be utilized to analyze results in collaboration with Dr. Harrison.

ELIGIBILITY:
Inclusion Criteria: (1) 18-28 years of age; (2) Currently matriculated undergraduate students at any university; and (3) Able to read, write, and speak in English

Exclusion Criteria: (1) Current regular meditation practice (>once/week); (2) Serious medical illness precluding regular class attendance; (3) Current substance abuse, suicidal ideation or eating disorder; and (4) History of bipolar or psychotic disorders or self-injurious behaviors.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

PRIMARY OUTCOMES:
Health Summary Score | Baseline, 3-month, 6-month
  The primary outcome is change in a college health summary score from baseline to 6 months follow-up, assessed using the following 7 evidence-based determinants of health relevant to college student well-being: body mass index; physical activity (MET minutes and step counts per week, using validated actigraphy and IPAQ); diet (mean daily fruit and vegetable consumption, utilizing validated food frequency questionnaire); alcohol consumption (mean drinks per day); sleep quantity (mean sleep hours per night); perceived stress (validated Perceived Stress Scale score); and loneliness (validated R-UCLA Loneliness Scale score). Secondary analyses will evaluate which of the seven domains are most driving associations. Further secondary analyses will determine if participant-identified health domains to focus on showed improvements in MB-College vs. control, restricting only to health domains identified by participants as having high readiness to change.

SECONDARY OUTCOMES:
Self-Awareness | Baseline, 3-month, 6-month
  Multidimensional Assessment of Interoceptive Awareness: 32-item measure
Attention Control | Baseline, 3-month, 6-month
  Sustained Attention to Response Task: a computerized go/no-go task that evaluates sustained attention, response inhibition as well as self-regulation.
Self-Compassion | Baseline, 3-month, 6-month
  Self-Compassion Scale- short form: 12 item version and evaluate both a total score as well as six sub-scales of self-compassion: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification.

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Loucks, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Personally de-identified data will be made available to researchers with IRB approval.

REFERENCES:
- [Derived] Nardi WR, Elshabassi N, Spas J, Zima A, Saadeh F, Loucks EB. Students experiences of an 8-week mindfulness-based intervention at a college of opportunity: a qualitative investigation of the mindfulness-based college program. BMC Public Health. 2022 Dec 13;22(1):2331. doi: 10.1186/s12889-022-14775-5. PMID 36514082
- [Derived] Nardi WR, Harrison A, Saadeh FB, Webb J, Wentz AE, Loucks EB. Mindfulness and cardiovascular health: Qualitative findings on mechanisms from the mindfulness-based blood pressure reduction (MB-BP) study. PLoS One. 2020 Sep 23;15(9):e0239533. doi: 10.1371/journal.pone.0239533. eCollection 2020. PMID 32966308
- [Derived] Loucks EB, Nardi WR, Gutman R, Saadeh FB, Li Y, Vago DR, Fiske LB, Spas JJ, Harrison A. Mindfulness-Based College: A Stage 1 Randomized Controlled Trial for University Student Well-Being. Psychosom Med. 2021 Jul-Aug 01;83(6):602-614. doi: 10.1097/PSY.0000000000000860. PMID 32947581